CLINICAL TRIAL: NCT06894927
Title: Hearing Screening in Adults Over 50 Years Old - Pilot Study
Brief Title: Hearing Screening in Adults Over 50 Years Old
Acronym: HSA50+
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Collaborators: The Society of General Practice, J. E. Purkyne Czech Medical Association (Unknown); Hospital Pardubice (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 202501 P01
Record Dates: First submitted 2025-01-02; First posted 2025-03-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-01

CONDITIONS: Hearing Loss, Bilateral Sensorineural, Progressive; Hearing Loss, Bilateral (Causes Other Than Tumors); Hearing Loss, Bilateral or Unilateral; Presbyacusis
Keywords: screening; hearing loss; adults; older; presbyacusis
MeSH Terms: conditions — Hearing Loss; Presbycusis | interventions — Audiometry, Pure-Tone; Acoustic Impedance Tests

STUDY DESIGN:
Intervention Model Description: single-arm quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): Participants over 50 years old.
  Interventions: Diagnostic Test: Screening HHIA questionnaire; Diagnostic Test: Whispered voice test; Diagnostic Test: Screening pure tone audiometry; Diagnostic Test: Pure Tone Audiometry; Diagnostic Test: Tympanometry

INTERVENTIONS:
Diagnostic Test: Screening HHIA questionnaire — Completion of the abbreviated (screening) version of the standardized "HHIA" questionnaire (Czech version).
Diagnostic Test: Whispered voice test — Whispered voice test conducted following the standardized protocol.
Diagnostic Test: Screening pure tone audiometry — Screening pure-tone audiometry at a level of 35 dB at the frequencies: 500, 1000, 2000, and 4000 Hz.
Diagnostic Test: Pure Tone Audiometry — Clinical Pure Tone Audiometry
Diagnostic Test: Tympanometry — Clinical Tympanometry

SUMMARY:
The goal of this single-arm quasi-experimental study is to evaluate the feasibility, effectiveness, and management of three different hearing screening methods in adults aged 50 years and older in the Czech Republic. The main questions it aims to answer are:

Are the selected hearing screening methods effective in detecting hearing loss in the target population? Can these methods be successfully implemented within the national healthcare system to address gaps in current practices?

Participants will:

1. Undergo hearing screening using all three methods, conducted by general practitioners, to assess their performance.
2. Complete follow-up evaluations conducted by ENT specialists to confirm diagnostic results.

DETAILED DESCRIPTION:
This single-arm quasi-experimental study involves a total of 330 participants aged 50 and older. The study evaluates the feasibility and effectiveness of three distinct hearing screening methods, conducted first by general practitioners and subsequently confirmed by ENT specialists, according to a standardized protocol.

Study Population and Interventions

Participants:

A total of 330 adults aged 50 years and older will be enrolled in the study.

Interventions:

The interventions are divided into two stages:

General Practitioners' Offices:

Before the screening:

Explanation of the screening process. Personal medical history review. Otoscopy and patient instruction.

Screening procedures (performed for all participants in the same order according to the standardized protocol):

1. Completion of the screening version of the standardized "HHIA" questionnaire (Czech version).
2. Whisper test conducted following the standardized protocol.
3. Screening pure tone audiometry performed according to the standardized protocol.

ENT Clinics:

Before the evaluation:

Explanation of the evaluation process. ENT-specific medical history review. Otoscopy and patient instruction.

Diagnostic procedures (performed for all participants in the same order according to the standardized protocol):

1. Pure tone audiometry conducted following the standardized protocol.
2. Tympanometry.

The findings will provide evidence for developing a comprehensive, national-scale hearing screening program for the aging population in the Czech Republic.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (IC) and consent for personal data processing (CPDP).
* Age 50 years or older.

Exclusion Criteria:

* Known diagnosed persistent hearing impairment.
* Inability to sufficiently understand study instructions due to language barriers.
* Medical condition preventing participation in all parts of the study.
* Inability or unwillingness to complete all parts of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Hearing Loss Detected by Pure-tone Screening Audiometry | From enrollment by the general practitioner to ENT examination, up to 4 weeks.
  This outcome measure evaluates the effectiveness of screening pure-tone audiometry at 35 dB at specific frequencies (500, 1000, 2000, and 4000 Hz) to detect hearing loss. Results will be compared to the reference standard (pure-tone audiometry performed at ENT clinics), calculating sensitivity, specificity, and agreement.
Number of Participants with Hearing Loss Detected by Whisper Test | From enrollment by the general practitioner to ENT examination, up to 4 weeks.
  This outcome measure assesses the effectiveness of the whispered voice test in detecting hearing loss. Results will be compared with the reference standard (pure-tone audiometry performed at ENT clinics), evaluating sensitivity, specificity, and overall agreement.
Number of Participants with Hearing Loss Detected by the HHIA Questionnaire | From enrollment by the general practitioner to ENT examination, up to 4 weeks.
  This outcome measure evaluates the effectiveness of the abbreviated Hearing Handicap Inventory for Adults (HHIA) questionnaire in identifying hearing loss. Results will be validated against the reference standard (pure-tone audiometry performed at ENT clinics), assessing sensitivity, specificity, and agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Chrobok, prof., M.D., CSc., Ph.D., Study Chair — University Hospital Hradec Kralove; MUDr. Michal Homoláč, Principal Investigator — University Hospital Hradec Kralove
Locations (2):
- Czechia (2):
  - University Hospital Hradec Kralove, Hradec Králové, Czech Republic
  - Pardubice Hospital, Pardubice, Czech Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WORLD HEALTH ORGANIZATION. Hearing Screening Considerations For Implementation. World Health Organization. 2021, 1-64.